CLINICAL TRIAL: NCT02934243
Title: Identification of Risk Factors Causing Difficulty in Laryngeal Mask Insertion
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Alessandro Di Filippo, Dr, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: GDSAIRWAY
Record Dates: First submitted 2016-10-13; First posted 2016-10-14 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2019-12

CONDITIONS: Anesthesia
Keywords: Laryngeal Masks; Ventilation; Risk factors
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- easy Laryngeal Mask insertion: patients in whom the insertion of the SIM has proven easy
  Interventions: Device: laryngeal mask insertion
- difficult Laryngeal Mask insertion: patients in whom the insertion of the SIM has proven difficult
  Interventions: Device: laryngeal mask insertion

INTERVENTIONS:
Device: laryngeal mask insertion — airway management with laryngeal mask

SUMMARY:
Even if the laryngeal mask (LM) is considered a very safe device with a low incidence of complications there may be situations where it is difficult to insert.

Therefore it seems appropriate to carry out a prospective observational study that will identify the risk factors relating to the positioning of LM for the purpose of identification and prediction of them.

From reading the literature and from the opinion of the experts with extensive practice in airway management (part of the Working Group "Management of Airway" of the Italian Society of Anaesthesia, Analgesia, Resuscitation and Intensive Care) some possible causes of difficulty in the insertion of laryngeal mask have been identified; these possible causes were listed in a report that will be distributed to the centers enrolled in the conduction of the study.

1,864 patients will be enrolled in 8 Italian research centers to calculate the relative risk of each of the factors analyzed in order to identify those that, in view of the LM positioning, must be modified to reduce the risk of failure and, secondly, to identify the risk factors whose presence may contraindicate the use of the device and indicate the use of alternative methods for airway management.

DETAILED DESCRIPTION:
Backgrounds Since its introduction into clinical practice in 1983, the laryngeal mask (LM) has found a role in the daily practice of anesthesiologists, including its use as a primary device in the airway management in both elective and emergency and as an emergency approach to the management of difficult airways.

Moreover, the insertion of the LM has become a common technique in the management of the airway, in particular outpatient surgery, where it is associated with a shorter recovery time, faster discharge and thus with a reduction of costs.

Even if the LM is considered a device very safe with a low incidence of complications, there may be situations where it is difficult to insert.

Aim of the study Some studies have concerned the causes that determine the difficulty in the insertion of an LM. They are retrospective studies and/or focused on the analysis of a single type of device.

Therefore, it seems appropriate to carry out a prospective observational study that will identify and weight the risk factors relating to the positioning of LM for the purpose of identification and prediction of them.

Methods From reading the literature and from the opinion of the experts with extensive practice in airway management (part of the Working Group "Management of Airway" of the Italian Society of Anaesthesia, Analgesia, Resuscitation and Intensive Care SIAARTI) some possible causes of difficulty in the insertion of laryngeal mask have been identified; these possible causes were listed in a report that will be distributed to the centers enrolled in the conduction of the study.

The centers will be selected based on the fact that between the researchers is including an anesthesiologist part of the Working Group "Airway management" of SIAARTI to act as supervisor.

Statistic Descriptive: for each quantitative variable will be reported mean, standard deviation, first and third quartiles, median, minimum and maximum. For each qualitative variable will be reported frequency and percentage of each category.

Explorative: The association between each risk factor and the proportion of incorrect insertion will be evaluated only in a univariate analysis, using the relative risk and its confidence interval.

Sample size: For a hypothesis test on the relative risk so specified H0: RR ≤ 1 H1: RR> 1 and considering an expected relative risk of 2, a proportion of 2.9% of the failures in the group of experts and a first type error equal to 5%, 832 patients per group are needed to ensure a power equal to 90%.

The limit of significance is set at 5%.

Expected results To calculate the relative risk of each of the factors analyzed in order to identify those that, in view of the LM positioning, can be modified to reduce the risk of failure and, secondly, to identify the risk factors whose presence may contraindicate the use of the device and indicate the use of alternative methods for airway management.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I-II
* Age between 18 and 65 years
* Airway management with laryngeal mask
* Signed informed consent to the study in the medical record

Exclusion Criteria:

* Diseases of the upper airways
* Risk of inhalation of gastric contents (previous gastric surgery, hiatal hernia, gastroesophageal reflux, peptic ulcer, stomach full, pregnancy)
* Large obese (BMI> 40)
* Sore throat, voice alteration
* A history of difficult intubation
* Intervention lasting more than 4 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients submitted to insertion of laryngeal mask collected in 8 Italian research centers
Sampling Method: Probability Sample
Enrollment: 432 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Success in the first attempt | Immediately after the attempt of insertion
  number

SECONDARY OUTCOMES:
Need for 2 or more attempts | Immediately after the attempt of insertion
  number
Substitution with another LM of different size | Immediately after the attempt of insertion
  number
Change in strategy (intubation, awakening) | Immediately after the attempt of insertion
  number
Ventilation difficulties | Immediately after the attempt of insertion
  number
Movement or swallowing after placement | Immediately after the attempt of insertion
  number

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Di Filippo, Dr, Principal Investigator — Azienda Ospedaliero-Universitaria Careggi
Locations (1):
- Alessandro Di Filippo, Florence, Italy

IPD SHARING:
Plan to Share IPD: Yes
All data collected were available for the researchers by direct information and divulgation by principal researcher
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: immediately and for the duration of the data collection
Access Criteria: email by principal researcher

REFERENCES:
- [Background] Brain AI. The laryngeal mask--a new concept in airway management. Br J Anaesth. 1983 Aug;55(8):801-5. doi: 10.1093/bja/55.8.801. PMID 6349667
- [Background] White PF. Ambulatory anesthesia advances into the new millennium. Anesth Analg. 2000 May;90(5):1234-5. doi: 10.1097/00000539-200005000-00047. No abstract available. PMID 10781489
- [Background] Suhitharan T, Teoh WH. Use of extraglottic airways in patients undergoing ambulatory laparoscopic surgery without the need for tracheal intubation. Saudi J Anaesth. 2013 Oct;7(4):436-41. doi: 10.4103/1658-354X.121081. PMID 24348297
- [Background] Brimacombe J. The advantages of the LMA over the tracheal tube or facemask: a meta-analysis. Can J Anaesth. 1995 Nov;42(11):1017-23. doi: 10.1007/BF03011075. PMID 8590490
- [Background] Apfelbaum JL, Hagberg CA, Caplan RA, Blitt CD, Connis RT, Nickinovich DG, Hagberg CA, Caplan RA, Benumof JL, Berry FA, Blitt CD, Bode RH, Cheney FW, Connis RT, Guidry OF, Nickinovich DG, Ovassapian A; American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Practice guidelines for management of the difficult airway: an updated report by the American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Anesthesiology. 2013 Feb;118(2):251-70. doi: 10.1097/ALN.0b013e31827773b2. No abstract available. PMID 23364566
- [Background] Berlac P, Hyldmo PK, Kongstad P, Kurola J, Nakstad AR, Sandberg M; Scandinavian Society for Anesthesiology and Intensive Care Medicine. Pre-hospital airway management: guidelines from a task force from the Scandinavian Society for Anaesthesiology and Intensive Care Medicine. Acta Anaesthesiol Scand. 2008 Aug;52(7):897-907. doi: 10.1111/j.1399-6576.2008.01673.x. PMID 18702752
- [Background] Apfelbaum JL, Walawander CA, Grasela TH, Wise P, McLeskey C, Roizen MF, Wetchler BV, Korttila K. Eliminating intensive postoperative care in same-day surgery patients using short-acting anesthetics. Anesthesiology. 2002 Jul;97(1):66-74. doi: 10.1097/00000542-200207000-00010. PMID 12131105
- [Background] Lubarsky DA. Fast track in the postanesthesia care unit: unlimited possibilities? J Clin Anesth. 1996 May;8(3 Suppl):70S-72S. doi: 10.1016/s0952-8180(96)90016-1. No abstract available. PMID 8695119
- [Background] Verghese C, Brimacombe JR. Survey of laryngeal mask airway usage in 11,910 patients: safety and efficacy for conventional and nonconventional usage. Anesth Analg. 1996 Jan;82(1):129-33. doi: 10.1097/00000539-199601000-00023. PMID 8712387
- [Background] Buckham M, Brooker M, Brimacombe J, Keller C. A comparison of the reinforced and standard laryngeal mask airway: ease of insertion and the influence of head and neck position on oropharyngeal leak pressure and intracuff pressure. Anaesth Intensive Care. 1999 Dec;27(6):628-31. doi: 10.1177/0310057X9902700612. PMID 10631418
- [Background] Katsiampoura AD, Killoran PV, Corso RM, Cai C, Hagberg CA, Cattano D. Laryngeal mask placement in a teaching institution: analysis of difficult placements. F1000Res. 2015 Apr 29;4:102. doi: 10.12688/f1000research.6415.1. eCollection 2015. PMID 26401265
- [Background] Ramachandran SK, Mathis MR, Tremper KK, Shanks AM, Kheterpal S. Predictors and clinical outcomes from failed Laryngeal Mask Airway Unique: a study of 15,795 patients. Anesthesiology. 2012 Jun;116(6):1217-26. doi: 10.1097/ALN.0b013e318255e6ab. PMID 22510864